CLINICAL TRIAL: NCT01062646
Title: A Randomized Controlled Trial of Multimodal Music Therapy for Children With Anxiety Disorders
Brief Title: Multimodal Music Therapy for Children With Anxiety Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Prof. Dr. Goldbeck, University Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUSICANXCHILD
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2010-02-04 (Estimated); Status verified 2006-05

CONDITIONS: Anxiety
Keywords: music therapy; multimodal psychotherapy; children; anxiety disorders; pediatric anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multimodal music therapy (Experimental): Multimodal music therapy comprises 16 sessions single music therapy, group music therapy (max. 6 children/group), parent-child sessions, and parent counseling. The manualized treatment integrates music therapy, behavioral interventions, and family-oriented interventions.
  Interventions: Behavioral: Multimodal music therapy
- community treatment as usual (Active Comparator)
  Interventions: Behavioral: Community treatment as usual

INTERVENTIONS:
Behavioral: Multimodal music therapy
  Arms: Multimodal music therapy
Behavioral: Community treatment as usual
  Arms: community treatment as usual

SUMMARY:
Multimodal music therapy (MT) for children ages 8 to 12 years with anxiety disorders is compared to community treatment as usual (TAU). 36 children were randomized either to MT or to TAU. Primary outcome is presence of an anxiety disorder at the end of treatment. Secondary outcomes are self- and parent-/teacher reported anxiety, co-morbid psychological symptoms, and quality of life. Stability of outcome is assessed six months after the end of treatment.

DETAILED DESCRIPTION:
Patients were enrolled in a community clinic and in an outpatient clinic for child and adolescent psychiatry/psychotherapy. Inclusion criteria: diagnosis of an anxiety disorder (separation anxiety disorder, general anxiety disorder, social phobia, specific phobia, or other anxiety disorder); age 8-12; no medication or stable medication during treatment; IQ>80; informed consent of caregivers and informed assent of patients. Outcome measures. Kiddie-SADS; STAIC-C, SPAIC, CDI; SDQ teacher report; CBCL 4-18; ILK quality of life inventory. Assessment time points: pre-intervention; post-intervention; 6-months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* age 8-12 years
* diagnosis of an anxiety disorder
* IQ>80
* informed consent and assent

Exclusion Criteria:

* anxiety disorder is not primary focus of treatment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Diagnosis of an anxiety disorder (DSM IV)

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Goldbeck, Ph.D., Principal Investigator — University Ulm